CLINICAL TRIAL: NCT04774159
Title: Low Dose ColchicinE in pAtients With Peripheral Artery DiseasE to Address Residual Vascular Risk: A Randomized Trial
Brief Title: Low Dose ColchicinE in pAtients With Peripheral Artery DiseasE to Address Residual Vascular Risk
Acronym: LEADER-PAD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Principal Investigator, Noel Chan, Principal Investigator, Population Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LEADER-PAD
Record Dates: First submitted 2021-02-21; First posted 2021-03-01 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-05

CONDITIONS: Peripheral Arterial Disease; Atherosclerosis of Extremities; Inflammation
Keywords: Acute limb ischemia; Myocardial Infarction; Stroke; Cardiovascular death; Mortality
MeSH Terms: conditions — Peripheral Arterial Disease; Inflammation; Myocardial Infarction; Stroke | interventions — Colchicine; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind and use of similarly active and placebo tablets.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colchicine (Active Comparator): Colchicine 0.5mg daily for the duration of the trial
  Interventions: Drug: Colchicine 0.5 MG Oral Tablet
- Colchicine-Placebo (Placebo Comparator): Colchicine-Placebo daily
  Interventions: Drug: Colchicine-Placebo

INTERVENTIONS:
Drug: Colchicine 0.5 MG Oral Tablet — Colchicine 0.5 mg tablet daily
  Active drug and placebo are of the same appearance and are indistinguishable. All investigators, study personnel and patients will be blinded to drug treatment assignment. Trial treatment supplies must be stored in a secure, limited-access location under the storage conditions specified on the IP supply label.
  Other Names: Colchicine
  Arms: Colchicine
Drug: Colchicine-Placebo — Colchicine-Placebo tablet
  Other Names: Colchicine-Placebo tablet
  Arms: Colchicine-Placebo

SUMMARY:
The Low dose ColchicinE in pAtients with peripheral Artery DiseasE to address residual vascular Risk (LEADER-PAD) trial will evaluate if anti-inflammatory therapy with colchicine will reduce vascular events in patients with symptomatic peripheral artery disease.

DETAILED DESCRIPTION:
The LEADER-PAD trial is a randomized, double blind, multicenter trial with an active run-in period, comparing low dose colchicine 0.5 mg daily with placebo in patients with symptomatic peripheral artery disease (PAD) to prevent vascular events (myocardial infarction, stroke, cardiovascular deaths, acute limb ischemia and vascular amputation). The sample size for the trial is 6,150 participants. The primary outcome for the trial is major adverse cardiovascular and limb events (MACE and MALE). This composite outcome consists of cardiovascular death, myocardial infarction, stroke and severe limb ischemia that requires a vascular intervention (i.e., pharmacological reperfusion, endovascular or surgical revascularization) or a major vascular amputation (defined as ankle/transtibial amputation or higher).

ELIGIBILITY:
Inclusion criteria:

1. Age > 18 years
2. Symptomatic atherosclerotic LE PAD fulfilling at least one of the following:

   a. Intermittent claudication with ankle/arm blood pressure ratio* (ABI ≤ 0.90) or artery stenosis ≥ 50% plus one of i. >1 vascular bed affected by atherosclerosis ii. Diabetes iii. Heart failure iv. Chronic kidney disease (eGFR < 60 mL/min/1.73 m2)

   b. Rest pain (mostly in foot) OR necrosis of limb OR gangrene of limb (corresponding to either Fontaine stages 3 or 4 OR Rutherford Classification categories 4 to 6). All must have an ankle/arm blood pressure ratio* (ABI ≤ 0.90) OR artery stenosis ≥ 50%.

   * In cases of incompressible ankle arteries, the presence of toe pressure ≤ 60 mm Hg or toe-brachial index ≤ 0.70 is acceptable

   c. Revascularization defined as limb bypass surgery or endovascular revascularization procedures (irrespective of the specific device used), including percutaneous transluminal angioplasty/stent of iliac or infra-inguinal arteries or extra-anatomical bypass surgery

   d. Leg or foot amputation for arterial vascular indications
3. Written or verbal informed consent from the patient

Exclusion Criteria:

1. Contraindication to colchicine
2. Long term requirement for colchicine for another clinical indication
3. Active diarrhoea
4. eGFR < 30 mL/min/1.73 m2
5. Cirrhosis or severe chronic liver disease
6. Woman who is pregnant, or breast-feeding or of child-bearing potential not protected by reliable contraception or is planning conception during the study
7. Current or planned long term use of cyclosporine, verapamil, HIV protease inhibitors, azole antifungals, or macrolide antibiotics (with the exception of azithromycin)
8. Patients who are deemed unlikely to return for follow-up
9. Patients with life expectancy < 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6150 (Estimated)
Dates: Start 2021-05-06 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular and limb events (MACE or MALE) | 3-5 years
  This composite outcome consists of cardiovascular deaths, myocardial infarction, stroke, and severe limb ischemia that requires a vascular intervention (i.e., pharmacological reperfusion, endovascular or surgical revascularization) or a major vascular amputation (defined as ankle/transtibial amputation or higher)

SECONDARY OUTCOMES:
Extended MALE | 3-5 years
  This composite outcome includes major adverse limb events (MALE) as well as revascularization for new or worsening claudication of new stenosis or occlusion detected on screening after a previous intervention
Cardiovascular death | 3-5 years
  Death will be classified as cardiovascular or non-cardiovascular. All deaths with a clear cardiovascular or unknown cause will be classified as cardiovascular. Only deaths due to a documented non-cardiovascular cause (e.g., cancer) will be classified as non-cardiovascular.
Myocardial infarction | 3-5 years
  Acute myocardial infarction (AMI) requires evidence of acute myocardial injury with clinical evidence of acute myocardial ischemia
Stroke | 3-5 years
  Stroke requires the presence of acute focal or global* neurological dysfunction caused by brain or retinal vascular injury due to primary hemorrhage or infarction.
Hospitalization | 3-5 years
  Admission to hospital for any reason
Acute or chronic limb-threatening ischemia | 3-5 years
  This is defined as an episode severe limb ischemia that requires an acute vascular intervention (i.e., pharmacological reperfusion, endovascular or surgical revascularization) or a major vascular amputation (defined as at ankle or transtibial amputation or higher).
All revascularization (coronary or cerebrovascular or lower limb or other peripheral revascularization) | 3-5 years
  Defined as coronary or cerebrovascular or lower limb or other peripheral revascularization
Total vascular amputation | 3-5 years
  All vascular amputations
Overall mortality | 3-5 years
  All cause (CV and non CV) deaths
Any thrombosis or thromboembolism (arterial and venous) | 3-5 years
  All arterial and venous thromboembolism
Fontaine Stage | 3-5 years
  This classification system grades the clinical presentation of patients to four stages of PAD
Standard Assessment of Global Everyday Activities (SAGEA) | 3-5 years
  The Standard Assessment of Global Everyday Activities (SAGEA) is a 15 item tool to assess activities of daily living including higher executive function used in social situations, everyday activities and basic activities of daily living. Scores range from 0 to 24 with higher scores indicating poorer function.It is a 15 items questionnaire and the scores will range from 0, describing a very independent participant over a broad spectrum of activities, to 48 describing a very dependent participant
Vascular Quality of Life Questionnaire-6 (VascQOL-6) | 3-5 years
  Six item vascular quality of life instrument: The total score is achieved by summarizing the score on each question, resulting in a score between 6 and 24. Higher value indicates better health status.
EuroQol 5 Dimension 5 Level (EQ-5D-5L) | 3-5 years
  A survey that measures quality of life across 5 domains. Each domain is scored on a 5-level severity ranking that ranges from "no problems" to "extreme problems".

OTHER OUTCOMES:
Occurrence of gastrointestinal toxicity (such as diarrhoea, nausea or vomiting) that results in study drug discontinuation | 3-5 years
  Safety outcome
Muscle pain (myalgia or myositis), that results in study drug discontinuation | 3-5 years
  Safety outcome
Infection (e.g., pneumonia) leading to hospitalization | 3-5 years
  Safety outcome
New diagnosis of cancer | 3-5 years
  Safety outcome
Renal insufficiency (defined as the need for dialysis or kidney transplant) | 3-5 years
  Other outcomes of interest
Neuropathy leading to study drug discontinuation | 3-5 years
  Other outcomes of interest
Neutropenia leading to study drug discontinuation | 3-5 years
  Other outcomes of interest
Bleeding | 3-5 years
  Other outcomes of interest

CONTACTS AND LOCATIONS:
Overall Officials: Noel C Chan, MD, Principal Investigator — Population Health Research Institute, Hamilton, Ontario, Canada
Locations (59):
- United States (17):
  - Yale School of Medicine, New Haven, Connecticut
  - University of Florida - Gainesville, Gainesville, Florida
  - Tampa General Hospital, Tampa, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Henry Ford Health System, Detroit, Michigan
  - Rutgers University, Newark, New Jersey
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke Regional Hospital, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Duke Raleigh Hospital, Raleigh, North Carolina
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Southwest Family Medicine, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Tech University Health Sciences, Lubbock, Texas
  - University of Washington Medical Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Universitair Ziekenhuis Leuven, Leuven, Belgium
- Brazil (10):
  - Clínica Procárdio, Blumenau, Santa Catarina
  - Sociedade Hospitalar Angelina Caron, Campina Grande do Sul
  - Hospital Universitário (CoraCentro Pesquisa Clinica), Canoas
  - Incore, Dois Vizinhos
  - Via Medica, Goiânia
  - Hospital Carlos Fernando Malzoni, Matão
  - Santa Casa de Misericórdia de Ponta Grossa, Ponta Grossa
  - Instituto de Cardiologia do Rio Grande do Sul, Porto Alegre
  - CPTEM - Centro de Pesquisa e Tecnologia Multidisciplinar, São Paulo
  - Hospital Alemão Oswaldo Cruz, São Paulo
- Canada (11):
  - University of Calgary, Peter Lougheed Centre Vascular Clinic, Calgary, Alberta
  - University of Alberta, Mazankowski Heart Institute, Edmonton, Alberta
  - Hamilton General Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Vascular Health Bronte, Oakville, Ontario
  - Corcare Cardiovascular Research Inc., Scarborough Village, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - CIUSSS du Nord-de-l'île-de-Montréal, Hôpital du Sacré-Cœur-de-Montréal, Montreal, Quebec
  - Centre intégré de santé et de services sociaux du Bas-Saint-Laurent, Rimouski, Quebec
- Ecuador (3):
  - Cardiolife, Quito, Pichincha
  - Hospital de Especialidades de las Fuerzas Armadas N 1, Quito, Pichincha
  - UniCarMeDr.D, Quito, Pichincha
- University Medical Center Utrecht, Utrecht, Netherlands
- Switzerland (5):
  - University Hospital Basel, Angiology, Basel
  - Ospedale Regionale Bellinzona e Valli - Ente Ospedaliero Cantonale, Bellinzona
  - HFR Fribourg, Fribourg
  - Hôpitaux Universitaires de Genève, Geneva
  - University Hospital Zurich, Clinic of Angiology, Zurich
- United Kingdom (11):
  - Royal Sussex County Hospital, Brighton, England
  - Southmead Hospital, Bristol, England
  - Kent and Canterbury Hospital, Canterbury, England
  - Derriford Hospital, Plymouth, England
  - Pinderfields Hospital, Wakefield, England
  - Royal Infirmary Edinburgh, Edinburgh, Scotland
  - Bradford Teaching Hospital, Bradford
  - Hull Royal Infirmary, Hull
  - The Leeds Teaching Hospital, Leeds
  - Glenfield Hospital, Leicester
  - St. George's University Hospitals, London

IPD SHARING:
Plan to Share IPD: No